CLINICAL TRIAL: NCT01588561
Title: Nicotine Related Brain Activity: The Influence of Smoking History and Blood Nicotine Levels, an Exploratory Study
Brief Title: Nicotine Related Brain Activity: The Influence of Smoking History and Blood Nicotine Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Scott Lukas, Director, McLean Imaging Center, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2005-p-001656; R01DA025065 (NIH)
Record Dates: First submitted 2012-04-06; First posted 2012-05-01 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-07

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous Nicotine (1.5 mg/70 kg) (Active Comparator): Participants are given a siingle infusion of nicotine (1.5 mg/70 kg), administered over 1 minute into the antecubital vein 10 minutes into their MRI scans
  Interventions: Drug: Intravenous Nicotine
- Saline - placebo (Placebo Comparator): Participants are given physiological saline, administered over 1 minute into the antecubital vein 10 minutes into their MRI scans
  Interventions: Other: Saline - placebo

INTERVENTIONS:
Drug: Intravenous Nicotine — Subjects received a single infusion of nicotine, 1.5 mg/70kg (New England Compounding Center, Framingham, MA), administered over 1 minute into the antecubital vein 10 minutes into their MRI scans.
  Other Names: IV Nicotine
  Arms: Intravenous Nicotine (1.5 mg/70 kg)
Other: Saline - placebo — Subjects received a single infusion of saline, administered over 1 minute into the antecubital vein 10 minutes into their MRI scans.
  Arms: Saline - placebo

SUMMARY:
In this study, we sought to explore brain activity in nicotine-dependent men in response to acute intravenous nicotine using pharmacological magnetic resonance imaging (phMRI).

DETAILED DESCRIPTION:
phMRI was used to evaluate brain activity in response to 1.5 mg/70 kg intravenous nicotine or saline. The nicotine and saline were administered on different visits. The time courses of individual subjects' nicotine levels were used as regressors to assess neural activity relating to the infusions. The influence of Smoking history and physiological measures on the response to nicotine were also investigated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 40 who currently smoke at least 15 cigarettes every day, and who fulfill DSM-IV diagnostic criteria for nicotine dependence will be eligible for participation.
* No evidence of clinically significant disease based upon complete medical history and physical examination by a qualified physician.
* Absence of DSM-IV Axis I Disorders other than nicotine dependence (305.10) as measured by the Structured Clinical Interview (SCID).
* Routine laboratory blood tests including complete blood count, electrolytes, BUN and creatinine, liver function tests, hepatitis panel and urinalysis will be performed. Laboratory parameters must be within the normal range. HBsAg must be negative but subjects who have hepatitis serology consistent with previous exposure to Hepatitis A, Hepatitis B, or Hepatitis C, but who do not have clinical and biochemical evidence of acute infection, will be acceptable.
* Hematocrit levels ≥ 39% for males and ≥ 35% for females.
* Serum pregnancy test (hCG beta subunit) results must be negative within 24 hrs of the study day.
* Normal ECG.
* A Body Mass Index (BMI-ratio of weight (W) to height (H) squared; W/H2=kg/m2) of between 18.0 and 27.0 for women and 21.4 to 29 for men.
* Subjects must be able to read and understand instructions, as well as provide a valid informed consent.

Exclusion Criteria:

* Participants with any lifetime DSM-IV Axis I disorder other than nicotine dependence.
* Participants with clinically significant medical disorders.
* Women who are pregnant as determined by laboratory testing for serum beta hCG.
* Women who use hormonal contraceptive medications will not be accepted, because this would confound the hormonal measures.
* Women with a mean BMI of outside the range 18.0-27.0 and men with a BMI outside the range 21.4-29.0.
* Participants with ferromagnetic implants or other contraindications to fMRI

  * Cardiac pacemakers
  * Metal clips on blood vessels (also called stents)
  * Artificial heart valves
  * Artificial arms, hands, legs, etc.
  * Brain stimulator devices
  * Implanted drug pumps
  * Ear implants
  * Eye implants or known metal fragments in eyes
  * Exposure to shrapnel or metal filings (wounded in military combat, sheet metal workers, welders, and others)
  * Other metallic surgical hardware in vital areas
  * Certain tattoos with metallic ink
  * Transdermal patches (eg. Orthro Evra, Nicoderm CQ)
  * Metal IUD (s)
* Participants who describe themselves as seeking treatment will not be selected but will be referred to local smoking cessation programs.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-10; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott E. Lukas, PhD, Principal Investigator — Mclean Hospital; Harrison G Pope, MD, Principal Investigator — Mclean Hospital
Locations (1):
- Alcohol and Drug Abuse Research Center at McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yamamoto RT, Rohan ML, Goletiani N, Olson D, Peltier M, Renshaw PF, Mello NK. Nicotine related brain activity: the influence of smoking history and blood nicotine levels, an exploratory study. Drug Alcohol Depend. 2013 Apr 1;129(1-2):137-44. doi: 10.1016/j.drugalcdep.2012.10.002. Epub 2012 Oct 29. PMID 23117126

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First, Then Nicotine: Placebo first, then Intravenous Nicotine (1.5 mg/70 kg)
- Nicotine First, Then Placebo: Intravenous Nicotine (1.5 mg/70 kg) first, then Placebo
Period: Overall Study
Arm/Group | Placebo First, Then Nicotine | Nicotine First, Then Placebo
Started | 14 | 1
First Injection (Visit 1) | 14 | 1
Rest Period (Generally 2-3 week rest period but a minimum of 1 month for women, based on menstrual cycles.) | 14 | 1
Second Injection (Visit 2) | 14 | 1
Completed | 14 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants. All participants were randomized to receive all interventions, so all participants are combined into one Arm/Group.
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 6
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 15
Pack-years [Mean (Standard Deviation); unit: pack-years] — calculated by reported daily cigarettes smoked divided by 20/pack and multiplied by the number of years reported smoking
  pack-years | 11.2 (10.5)
Fagerström score [Mean (Standard Deviation); unit: units on a scale] — Fagerstrom test for nicotine dependence:
  http://ndri.curtin.edu.au/btitp/documents/Fagerstrom_test.pdf Scores ranged between 1 to 10, 1-2 = low dependence, 3-4 = low to moderate dependence, 5-7 = moderate dependence, 8+ = high dependence
  units on a scale | 6.0 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Peak Nicotine Levels
Description: Peak nicotine level in each participant
Time Frame: 0, 2, 4, 6, 8, 10, 12, 14, 16, 20, 30 minutes post-infusion
Population: Peak nicotine levels were only measured during the nicotine study intervention. One participant had incomplete serum nicotine results and was not included.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Nicotine: Intravenous Nicotine (1.5 mg/70 kg)
- Placebo: Saline infusion
Arm/Group | Nicotine | Placebo
Number analyzed (Participants) | 14 | 14
ng/ml | 16.1 (8) | 0 (0)

2. Primary Outcome: Number of Brain Regions With a Change in Brain Activity Relative to Saline
Description: PhMRI analysis of the differential response of nicotine compared to the saline condition when analyzed with the nicotine time course.
  The main dependent variable in this study, Blood Oxygen Level Dependent (BOLD) measures of brain activity (via fMRI) data does not exist in a vacuum-it is always relative to another measure of brain activity, typically collected at rest or after a placebo injection. So we collected the data after the IV placebo injection alone and the IV nicotine injection alone, but then need applied mathematical CONTRASTS to the data. This procedure results in the brain activity maps.
Time Frame: 40 minutes after infusion
Population: The data from three subjects were not included in the imaging results, one due to incomplete serum nicotine results, one due to a misalignment of the head in the scanner, which resulted in incomplete brain coverage, and one subject had a combination of excessive motion and abnormal anatomy.
Measure: Number; unit: brain regions
Arm/Group | Nicotine
Number analyzed (Participants) | 12
brain regions
  Increased BOLD Signal | 9
  Decreased BOLD Signal | 5
Statistical Analysis 1: Comparison: Nicotine; Test type: Other; Increased signal: Insula, Putamen, Cingulate, Paracingulate, Calcarine cortex, Lingual gyrus, Frontal pole, Fusiform gyrus, Cerebellum. Decreased signal:Thalamus, Temporal gyri, Hippocampus (left), Caudate, Cerebellum

3. Secondary Outcome: Number of Brain Regions With a Change in Brain Activity Relative to Saline When Analyzed With the Nicotine Time Course Controlling for Smoking History
Description: PhMRI analysis of the differential response of nicotine compared to the saline condition when analyzed with the nicotine time course controlling for smoking history (pack years).
  The main dependent variable in this study, Blood Oxygen Level Dependent (BOLD) measures of brain activity (via fMRI) data does not exist in a vacuum-it is always relative to another measure of brain activity, typically collected at rest or after a placebo injection. So we collected the data after the IV placebo injection alone and the IV nicotine injection alone, but then need applied mathematical CONTRASTS to the data. This procedure results in the brain activity maps.
Time Frame: 40 minutes after infusion
Population: as for outcome 2
Measure: Number; unit: brain regions
Arm/Group | Nicotine
Number analyzed (Participants) | 12
brain regions
  Increased BOLD Signal | 9
  Decreased BOLD Signal | 4
Statistical Analysis 1: Comparison: Nicotine; Test type: Other; Increased signal: Insula, Putamen, Pallidum, Cingulate, Thalamus, Operculum, OBF cortex, Lingual gyrus, Cerebellum. Decreased signal: Hippocampus (left), Parahippocampus (left), Caudate, Cerebellum

4. Secondary Outcome: Number of Brain Regions With a Change in Brain Activity Relative to Saline When Analyzed With Smoking History Controlling for Nicotine
Description: PhMRI analysis of the differential response of nicotine compared to the saline condition when analyzed with smoking history (pack years) controlling for nicotine. The main dependent variable in this study, Blood Oxygen Level Dependent (BOLD) measures of brain activity (via fMRI) data does not exist in a vacuum-it is always relative to another measure of brain activity, typically collected at rest or after a placebo injection. So we collected the data after the IV placebo injection alone and the IV nicotine injection alone, but then need applied mathematical CONTRASTS to the data. This procedure results in the brain activity maps.
Time Frame: 40 minutes after infusion
Population: as for outcome 2
Measure: Number; unit: brain regions
Arm/Group | Nicotine
Number analyzed (Participants) | 12
brain regions
  Increased BOLD Signal | 9
  Decreased BOLD Signal | 7
Statistical Analysis 1: Comparison: Nicotine; Test type: Other; Increased signal: Insula (bilateral), Cingulate, Pretcentralgyrus, Thalamus (bilateral), Putamen (bilateral), Pallidum (bilateral), Amygdala (bilateral), Ventral tegmental area, Accumbens Nuclei. Decreased signal: Insula (left inferior), OBF cortex, Frontal&Temporal poles, Hippocampus (bilateral), Parahippocampus (bilateral), Accumbens nuclei, Cerebellum

5. Secondary Outcome: Final Nicotine Levels
Description: Final nicotine level in each participant
Time Frame: 30 minutes post-infusion
Population: One participant had incomplete serum nicotine results and was not included.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Nicotine | Placebo
Number analyzed (Participants) | 14 | 14
ng/ml | 8.2 (2.2) | 0 (0)

ADVERSE EVENTS:
Groups:
- Nicotine: Nicotine infusion
- Saline: Saline infusion
Arm/Group | Nicotine | Saline
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 2/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine (N=15) | Saline (N=15)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Transient tightness in chest (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small number of subjects completed due to a large shortage of Nicotine Bitartrate (the chemical used to create our IV Nicotine). We were unable to receive new nicotine shipments from 4/14 -2/15.Without this nicotine it was impossible to run subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes